CLINICAL TRIAL: NCT00777244
Title: Efficacy of Adjuvant Mitotane Treatment in Prolonging Recurrence-free Survival in Patients With Adrenocortical Carcinoma at Low-intermediate Risk of Recurrence
Brief Title: Efficacy of Adjuvant Mitotane Treatment (ADIUVO)
Acronym: ADIUVO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Alfredo Berruti, Prof., University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2007-007262-38
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Adrenocortical Carcinoma
Keywords: mitotane; adjuvant therapy; disease free survival
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — Mitotane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Follow-up (No Intervention): Arm B
- Mitotane (Experimental): Arm A
  Interventions: Drug: MITOTANE

INTERVENTIONS:
Drug: MITOTANE — mitotane will be administered at a starting dose of 1.5 g/day and increased in case of good gastrointestinal tolerance on day 2 to 3 g/day, on day 3 to 4.5 g/day, and on day 4 to 6 g/day. A dose of 6 g/day will be administered until first mitotane blood level is assessed. Further adjustment of dosage will be performed according to blood concentrations and tolerability.
  Other Names: Mitotane (Lysodren)
  Arms: Mitotane

SUMMARY:
Study Rationale Adrenocortical carcinoma (ACC) is a very rare disease with a high risk of relapse after radical surgery. The efficacy of adjuvant mitotane treatment is suggested by a retrospective multicenter international study showing that postoperative mitotane treatment was associated with a significant reduction of the risk of relapse and death. However, these promising results need confirmation in a randomized prospective study. Caution should be adopted particularly in patients with low risk of disease relapse, in whom the benefit of therapy should be weighted against the side effects. Even if an adjuvant treatment seems justified in patients at high risk of relapse, a randomised prospective study is needed to assess whether such a treatment is efficacious in patients at low-intermediate risk.

The purpose of the present study is to determine whether adjuvant mitotane treatment is effective in prolonging the disease free survival in patients with adrenocortical carcinoma at low-intermediate risk of progression who underwent radical resection

DETAILED DESCRIPTION:
Endpoints Primary : To compare DFS (Disease Free Survival), defined as the time between the date of randomization until documentation of any of the following failures (whichever occurs first): -local or distant recurrence of disease;-death from any cause or completion of follow-up.

Secondary:

To compare OS (Overall Survival), defined as the time interval between the date of randomization and the date of death from any cause or the last known alive date;· To compare quality of life measured by EORTC-QLQ-C30· To compare toxicity, graded according to the NCI-CTG criteria;· To compare DFS and OS in patients who achieve or not serum mitotane concentrations > 14 mg/L;· To compare DFS and OS between the 2 arms in patients subgroups stratified according to: type of hormone secretion, stage of disease, histopathologic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of ACC according to Weiss system by a national reference pathologist who has to be nominated before study initiation.
* Low-intermediate risk of relapse defined as:

  * Stage I-III (according to ENSAT classification 2008; see Appendix 2)
  * Microscopically complete resection, defined as no evidence of microscopic residual disease based on surgical reports, histopathology and post-operative imaging. Detailed pathological and surgical reports prepared according to guidelines detailed in appendix x and y should be available for assessment.
  * Ki 67 < 10%
* Post-operative imaging (thoracic and whole abdominal CT with contrast medium or MRI) demonstrating no evidence of disease within 4 weeks from randomization
* Age > 18 years
* ECOG performance status 0-2 (Appendix 3)
* Adequate bone marrow reserve (neutrophils > 1000/mm3 and platelets > 80000/ mm3)
* Ability to comply with the protocol procedures (including geographic accessibility)
* Written informed consent

Exclusion Criteria:

* Time between primary surgery and randomization > 3 months.
* Repeat surgery for recurrence of disease
* Presence of autonomous adrenocortical hormone secretion despite the absence of disease detectable with imaging techniques
* History of prior malignancy, except for cured non-melanoma skin cancer, cured in situ cervical carcinoma, or other treated malignancies with no evidence of disease for at least three years
* Renal insufficiency (creatinine clearance < 40 ml/min) or liver insufficiency (serum bilirubin > 2 times the upper normal range and/or serum transaminases (AST/SGOT, ALT/SGPT, but not gamma Glutamyl Transpeptidase) >3 times the upper normal range). Creatinine clearance may be calculated according to validated formulas (Crockoft's or MDRD)
* Pregnancy or breast feeding
* Previous or current treatment with mitotane or other antineoplastic drugs for ACC
* Previous radiotherapy of the tumor bed (for ACC).
* Any other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-04; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Disease Free survival | Till the last follow up
  Survival in years

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Terzolo, MD, Study Chair — Internal Medicine, Department of Clinical and Biological Sciences, University of Turin, Italy; Martin Fassnacht, MD, Study Director — Department of Internal Medicine, University of Wuerzburg, Germany; Alfredo Berruti, MD, Study Chair — Medical Oncology, Department of Clinical and Biological Sciences, University of Turin; Eric Baudin, MD, Principal Investigator — Oncologie Endocrinienne et Médecine Nucléaire, Institut Gustave Roussy, Villejuif, France.; Harm Haak, MD, Principal Investigator — Department of Internal Medicine, Máxima Medical Centre, Eindhoven, The Netherlands
Locations (28):
- United States (2):
  - Medical Oncology Branch - Center for Cancer Research - National Cancer Institute, Bethesda, Maryland
  - Endocrine Oncology - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
- Endocrinologie - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Canada
- France (6):
  - Endocrinologie - CHU Besançon Hôpital Jean Minjoz, Besançon
  - Endocrinologie - CHU Lyon Hôpital Pierre Wertheimer, Bron
  - Endocrinologie - Hôpital A. Michallon, La Tronche
  - Endocrinologie - Cochin, APHP, Paris
  - Endocrinologie - CHU Toulouse Hôpital Larrey, Toulouse
  - Endocrinologie - Institut de Cancérologie Gustave Roussy, Villejuif
- Germany (6):
  - University Hospital Campus Mitte Charitè, Berlin, Berlin
  - University Hospital of Dresden, Dresden
  - University Hospital of Düsseldorf, Düsseldorf
  - Center for Endocrine Tumors - ENDOC, Hamburg
  - University Medicin Centre of Munchen, München
  - University Hospital Wuerzburg, Endocrinology, Würzburg
- Italy (11):
  - A.O.Universitaria Arcispedale S.Anna Ferrara, Ferrara, Fe
  - UO Oncologia Medica - AO Spedali Civili, Brescia
  - Università degli studi di Firenze, Florence
  - Azienda Ospedaliera di Foggia, Foggia
  - Ospedale Cà Granda-Niguarda-Milano, Milan
  - Azienda Ospedaliera San Luigi, Orbassano
  - Department of Clinical and Biological Sciences, University of Turin, Internal Medicine 1, Orbassano
  - Azienda Ospedaliera Padova, Padua
  - Università degli studi di Palermo, Palermo
  - Policlinico Universitario A. Gemelli, Roma
  - A.O.U. San Giovanni Battista - Molinette, Torino
- Dept. of Internal Medicine Maxima Medisch Centrum, Eindhoven, Netherlands
- Cancer Research UK Clinical Trials Unit (CRCTU) - School of Cancer Sciences - University of Birmingham, Birmingham, Edgbaston, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Terzolo M, Angeli A, Fassnacht M, Daffara F, Tauchmanova L, Conton PA, Rossetto R, Buci L, Sperone P, Grossrubatscher E, Reimondo G, Bollito E, Papotti M, Saeger W, Hahner S, Koschker AC, Arvat E, Ambrosi B, Loli P, Lombardi G, Mannelli M, Bruzzi P, Mantero F, Allolio B, Dogliotti L, Berruti A. Adjuvant mitotane treatment for adrenocortical carcinoma. N Engl J Med. 2007 Jun 7;356(23):2372-80. doi: 10.1056/NEJMoa063360. PMID 17554118
- [Derived] Terzolo M, Fassnacht M, Perotti P, Libe R, Kastelan D, Lacroix A, Arlt W, Haak HR, Loli P, Decoudier B, Lasolle H, Quinkler M, Haissaguerre M, Chabre O, Caron P, Stigliano A, Giordano R, Zatelli MC, Bancos I, Fragoso MCBV, Canu L, Luconi M, Puglisi S, Basile V, Reimondo G, Kroiss M, Megerle F, Hahner S, Kimpel O, Dusek T, Nolting S, Bourdeau I, Chortis V, Ettaieb MH, Cosentini D, Grisanti S, Baudin E, Berchialla P, Bovis F, Sormani MP, Bruzzi P, Beuschlein F, Bertherat J, Berruti A. Adjuvant mitotane versus surveillance in low-grade, localised adrenocortical carcinoma (ADIUVO): an international, multicentre, open-label, randomised, phase 3 trial and observational study. Lancet Diabetes Endocrinol. 2023 Oct;11(10):720-730. doi: 10.1016/S2213-8587(23)00193-6. Epub 2023 Aug 21. PMID 37619579
- See also: study website — https://www.epiclin.it/adiuvo